CLINICAL TRIAL: NCT03996382
Title: Prevalence of Wild Type Transthyretin Cardiac Amyloidosis in Patients Operated for Idiopathic Carpal Tunnel Syndrome
Acronym: CACTuS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Steen Hvitfeldt Poulsen, Professor, Aarhus University Hospital Skejby
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-330-18
Record Dates: First submitted 2019-06-17; First posted 2019-06-24 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Amyloidosis Cardiac; Carpal Tunnel Syndrome
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspicion of cardiac amyloidosis (Other): Patients who display signs of cardiac amyloidosis will be referred for further diagnosis.
  Interventions: Diagnostic Test: DPD Scintigraphy

INTERVENTIONS:
Diagnostic Test: DPD Scintigraphy — Confirms/Refutes diagnosis of cardiac amyloidosis.

SUMMARY:
Wild-type transthyretin cardiac amyloidosis is an underdiagnosed depository disease in which fibril monomers of misfolded amyloid protein accumulates in various tissues, including the heart, and cause tissue dysfunction.

Before onset of cardiac symptoms, many patients will have undergone surgery for idiopathic carpal tunnel syndrome since the protein also deposits in the transversal carpal ligament of the hand.

This study investigates patients previously operated for idiopathic carpal tunnel syndrome to determine if they display signs and symptoms of cardiac amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients above sixty years of age previously operated for idiopathic carpal tunnel syndrome within the Region of Central Denmark (Region Midtjylland) the last five years.
* Informed written and verbal consent

Exclusion Criteria:

* Operation by different indication such as

  * Fracture
  * Ganglion
  * Tumors
  * Osteophytes
  * Rheumatoid Arthritis
  * Persistent medial artery
  * Metabolic causes
* Alcoholism
* Hyperthyroidism
* Myxedema

  * Hereditary Cardiac Amyloidosis
  * Known WT ATTR
  * AL Amyloidosis
  * Myelomatosis
  * MGUS and Morbus Waldenström

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of cardiac amyloidosis. | Through study completion, an average of 2 years.
  The prevalence of cardiac amyloidosis among patients previously operated for ipiopathic carpal tunnel syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Heart Disease, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided